CLINICAL TRIAL: NCT05641896
Title: A Phase 2, Multicenter, Single Arm, Open Label, Non-Randomized Study of [18F]FAPI-74 PET in Patients With Gastrointestinal Cancers
Brief Title: Study of [18F]FAPI-74 PET in Patients With Gastrointestinal Cancers
Acronym: 18F-FAPI-74 GI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOFIE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18FFAPI-2023P2
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Cancers; Cholangiocarcinoma; Gastric Cancer; Colorectal Cancer; Pancreatic Ductal Adenocarcinoma; Hepatocellular Carcinoma
Keywords: Fibroblast Activation Protein; Fibroblast Activation Protein Inhibitor; FAPI; Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Cholangiocarcinoma; Stomach Neoplasms; Colorectal Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]FAPI-74 PET/CT (Experimental): Patients receive [18F]FAPI-74 intravenously followed by PET/CT 60 minutes (+/-10minutes) later
  Interventions: Drug: [18F]FAPI-74 PET/CT

INTERVENTIONS:
Drug: [18F]FAPI-74 PET/CT — [18F]FAPI-74 is a radioactive diagnostic agent indicated for use with Positron Emission Tomography (PET) imaging for the detection of Fibroblast Activation Protein (FAP) positive cancer cells and cancer-associated fibroblasts (CAF) in patients with gastrointestinal cancers.

SUMMARY:
Prospective, multi-center, open label, non-randomized clinical trial to assess efficacy of [18F]FAPI-74 to detect FAP expressing cells in patients diagnosed with gastrointestinal cancers, including hepatocellular carcinoma, cholangiocarcinoma, gastric, pancreatic and colorectal cancer. The [18F]FAPI-74 PET scan will be acquired in patients with proven GI cancers after initial staging using institutional standard methods. The PET scan results will be compared to FAP immunohistochemistry (as the primary objective) and histopathology (as the secondary objective) of the biopsied or resected tissues.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of gastrointestinal (GI) malignancy, including hepatocellular carcinoma, cholangiocarcinoma, gastric, pancreatic and colorectal cancer
* Available tissue sample obtained through biopsy or to be obtained through scheduled biopsy and/or surgical resection
* No treatment received between tissue sample taken and [18F]FAPI-74 PET
* Anatomic imaging (e.g., CT, MRI) obtained within ≤ 28 days of consent
* Age ≥ 18 years
* Completed informed consent as determined per the IRB of record

Exclusion Criteria:

* Pregnant as determined by a pregnancy test as per institutional guidelines for individuals of child-bearing potential
* Declining to use effective contraceptive methods during the study (for individuals of child-producing potential)
* Need for emergent surgery that would be delayed by participation
* Bacterial, viral, or fungal infections requiring systemic therapy, that are expected to impact FAP expression in the opinion of the sponsor or their designee
* Serious co-morbidities and serious nonmalignant disease (e.g., hydronephrosis, kidney failure, liver failure, systemic or local inflammatory or autoimmune diseases or other conditions) that in the opinion of the investigator, physician of record and/or Sofie could compromise subject safety and/or protocol objectives
* Known diagnosis of an autoimmune disorder that is expected to impact FAP expression in the opinion of the sponsor or their designee
* Patients receiving any other investigational agent within the past 28 days
* Breastfeeding. Note: nursing parents are allowed if the potential participant commits to pumping breast milk and discarding it from injection to ≥ 24 hours from the time of the [18F]FAPI-74 injection
* Known hypersensitivity to any excipients used in [18F]FAPI-74: trace amounts of sodium acetate, sodium ascorbate, ascorbic acid, ethanol, acetonitrile or AlCl.
* Renal or liver function impairment* *Defined by liver impairments as AST>3x the upper limit of normal, ALT>3x the upper limit of normal, or bilirubin>1.5x the upper limit of normal. Renal impairment as defined by a creatinine clearance of >1.5x the upper limit of normal utilizing the Cockcroft Gault formula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Positive predictive value will be determined on a per-lesion basis for all lesions with tissue available for FAP analysis. | Through study completion, 2 years
  Lesions positive for FAP as detected by immunohistochemistry and Lesions positive for FAP as detected by [18F]FAPI-74 PET imaging

SECONDARY OUTCOMES:
Positive predictive value will be determined on a per-lesion basis for all lesions with tissue available for histopathology. | Through study completion, 2 years
  Malignant lesions as detected by histopathology and Lesions positive for FAP as detected by [18F]FAPI-74 PET imaging
Further characterize the safety profile of [18F]FAPI-74 in subjects utilizing Common Terminology Criteria for Adverse Events (CTCAE v5) | Through study completion, 2 years
  Incidence and severity of treatment emergent adverse events occurring within 24 hours.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California Los Angeles (UCLA) Health, Los Angeles, California
  - Massachusetts general hospital, Boston, Massachusetts
  - BAMF Health, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Northwell Health, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York

IPD SHARING:
Plan to Share IPD: Undecided